CLINICAL TRIAL: NCT04411797
Title: Impact of Stigma in Siblings of Young Patients With Schizophrenic Disorders
Acronym: STIG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Januel (Other)
Responsible Party: Sponsor-Investigator, Januel, Head of clinical research unit, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Other Study IDs: 10477M-STIG
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: The Impact of Stigma on the Quality of Life of People With Schizophrenic Disorders and Their Siblings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impact of stigma on the empathy and quality of life of people with schizophrenic disorders and their siblings.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Person with Schizophrenic Disorder

1. Aged between 18 and 35.
2. Medical follow-up in progress
3. DSM-5 diagnosis of Schizophrenia Spectrum Disorder
4. Reading and understanding the information and non-opposition form
5. Person affiliated to a social protection scheme or beneficiary of State Medical Aid
6. Volunteer mastering the French language

Exclusion Criteria:

Non-inclusion criteria for the person with schizophrenic disorders:

1. Clinical condition incompatible with testing 2. Current or less than one month's commitment to another research protocol 3. A person who is subject to a safeguard measure of justice 4 A person of full age under guardianship 5. Minor patients with mental disorders 6. Pregnant or breastfeeding women Version 1.2 date 19-05-2020 7. A person in situations of social fragility (persons deprived of liberty by a judicial or administrative decision, hospitalized persons) 8. Persons incapable or unable to give consent

Inclusion Criteria:

Inclusion criteria for a sibling member:

1. Age of 16 years or older
2. Volunteer with a sibling included in the study with a diagnosis of schizophrenia according to DSM-5.
3. Reading and understanding the information and non-opposition form
4. Volunteer affiliated to a social protection scheme or beneficiary of State Medical Aid
5. Volunteer mastering the French language

Criteria for non-inclusion of siblings:

1. Clinical condition incompatible with testing
2. Current or less than one month's commitment to another research protocol
3. Brother or sister subject to a measure of safeguard of justice 4 Brother or sister under curatorship

5. Brother or sister with mental health problems 6. Minor siblings under 16 years of age 7. A pregnant or nursing sister 8. Brother or sister in situations of social fragility (Persons deprived of liberty by a judicial or administrative decision, hospitalized persons) 9.Brother or sister incapable or unable to give consent

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: people with schizophrenic disorders and the subjective sense of stigma and siblings of people with schizophrenic disorders
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-12-25 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
Internalized Stigma of Mental Illness Scale | 1 hour and half
  for people with schizophrenic disorders

CONTACTS AND LOCATIONS:
Overall Officials: Davtian Hélène, Doctor, Principal Investigator — Les Funambules - Falret